CLINICAL TRIAL: NCT01917552
Title: Phase III Study of Adjuvant Capecitabine vs Observation Alone in Curatively Resected Stage IB (by AJCC 6th Edition) Gastric Cancer(KCSG ST14-05)
Brief Title: Adjuvant Capecitabine Versus Observation Alone in Curatively Resected Stage IB Gastric Cancer((KCSG ST14-05): CATALYSIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Ulsan University Hospital (Other); Seoul National University Bundang Hospital (Other); Gangnam Severance Hospital (Other); Seoul National University Boramae Hospital (Other); Ajou University School of Medicine (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Hallym University Medical Center (Other); Inje University Haeundae Paik Hospital (Other); Kyung Hee University Hospital (Other); Gachon University Gil Medical Center (Other); Kangbuk Samsung Hospital (Other); Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Min-Hee Ryu, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC1301
Record Dates: First submitted 2013-07-30; First posted 2013-08-06 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer
Keywords: Gastric adenocarcinoma, gastroesophageal junction adenocarcinoma, adjuvant, capecitabine, gastric cancer, stage 1b
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- capecitabine (Experimental): capecitabine 1250 milligram (mg) / m² po bid (D1-14)
  Interventions: Drug: capecitabine
- observation (No Intervention)

INTERVENTIONS:
Drug: capecitabine — capecitabine 1250 milligram (mg) / m² po bid (D1-14)
  Other Names: Xeloda
  Arms: capecitabine

SUMMARY:
multi-center, prospective, randomized, open-label phase III

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label phase III study of adjuvant chemotherapy after curative resection in patients with pathologic stage IB (by AJCC 6th edition) gastric cancer with at least one additional risk factor (additional risk factors for recurrence include age >65 years, male gender, presence of lymphovascular invasion, presence of perineural invasion). The superiority design will compare the efficacy and safety profiles of adjuvant capecitabine (Arm A) versus observation alone (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Curatively resected gastric or gastroesophageal junction adenocarcinoma
* Pathologic stage IB (by AJCC 6th edition) with at least one additional risk factor for recurrence (additional risk factors for recurrence include age >65 years, male gender, presence of lymphovascular invasion, presence of perineural invasion).
* Age: 18 -74years
* ECOG performance status: 0-2
* Adequate bone marrow function (ANC >1,500/uL, Platelets 100,000/uL, and Hb > 8.0 g/dL)
* Adequate renal function (serum creatinine < 1.5 mg/dL)
* Adequate hepatic function (bilirubin < 1.5 mg/dL, ALT and AST < 3 times upper limit of normal)
* Written informed consent

Exclusion Criteria:

* Pregnant or lactating women.
* Women of childbearing potential with either a positive pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-child bearing potential.
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study medication and until 3 months after discontinuation of the study medication.
* Any evidence of metastatic disease (including presence of tumor cells in the ascites).
* Previous chemotherapy or radiotherapy for the currently treated gastric cancer.
* No recovery from serious complications of gastrectomy.
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake.
* Clinically significant (i.e. active) cardiac disease: e.g. unstable angina, symptomatic coronary artery disease, New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication or myocardial infarction within the last 6 months.
* Lack of physical integrity of the upper gastrointestinal tract or those who have malabsorption syndrome likely to influence absorption of capecitabine, or inability to take oral medication.
* Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease.
* Organ allografts requiring immunosuppressive therapy.
* Received any investigational drug or agent/procedure, i.e. participation in another trial within 4 weeks before randomization.
* Requirement for concurrent use of the antiviral agent sorivudine (antiviral) or chemically related analogues, such as brivudine.
* Positive serologic test for HIV

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2013-08-19 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival | 8 years
  To demonstrate that capecitabine is superior to observation only (control arm) in terms of recurrence-free survival in curatively resected stage IB gastric cancer.

SECONDARY OUTCOMES:
overall survival | 8 years
  To compare overall survival in the capecitabine arm compared with the control arm.
Safety profiles | 8years
  Toxicity profiles will be assessed with the patient 28 +/- 3 days after the last intake of study medication is required. (treatment arm only)

CONTACTS AND LOCATIONS:
Overall Officials: Min-Hee Ryu, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

REFERENCES:
- [Background] Ajani JA, Faust J, Ikeda K, Yao JC, Anbe H, Carr KL, Houghton M, Urrea P. Phase I pharmacokinetic study of S-1 plus cisplatin in patients with advanced gastric carcinoma. J Clin Oncol. 2005 Oct 1;23(28):6957-65. doi: 10.1200/JCO.2005.01.917. Epub 2005 Sep 6. PMID 16145066
- [Background] Bang YJ, Kim YW, Yang HK, Chung HC, Park YK, Lee KH, Lee KW, Kim YH, Noh SI, Cho JY, Mok YJ, Kim YH, Ji J, Yeh TS, Button P, Sirzen F, Noh SH; CLASSIC trial investigators. Adjuvant capecitabine and oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): a phase 3 open-label, randomised controlled trial. Lancet. 2012 Jan 28;379(9813):315-21. doi: 10.1016/S0140-6736(11)61873-4. Epub 2012 Jan 7. PMID 22226517
- [Background] Diasio RB. Sorivudine and 5-fluorouracil; a clinically significant drug-drug interaction due to inhibition of dihydropyrimidine dehydrogenase. Br J Clin Pharmacol. 1998 Jul;46(1):1-4. doi: 10.1046/j.1365-2125.1998.00050.x. PMID 9690942
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Kang YK, Lee SS, Yoon DH, Lee SY, Chun YJ, Kim MS, Ryu MH, Chang HM, Lee JL, Kim TW. Pyridoxine is not effective to prevent hand-foot syndrome associated with capecitabine therapy: results of a randomized, double-blind, placebo-controlled study. J Clin Oncol. 2010 Aug 20;28(24):3824-9. doi: 10.1200/JCO.2010.29.1807. Epub 2010 Jul 12. PMID 20625131
- [Background] Kolesar JM, Johnson CL, Freeberg BL, Berlin JD, Schiller JH. Warfarin-5-FU interaction--a consecutive case series. Pharmacotherapy. 1999 Dec;19(12):1445-9. doi: 10.1592/phco.19.18.1445.30897. PMID 10600095
- [Background] Lee JL, Kang YK, Kang HJ, Lee KH, Zang DY, Ryoo BY, Kim JG, Park SR, Kang WK, Shin DB, Ryu MH, Chang HM, Kim TW, Baek JH, Min YJ. A randomised multicentre phase II trial of capecitabine vs S-1 as first-line treatment in elderly patients with metastatic or recurrent unresectable gastric cancer. Br J Cancer. 2008 Aug 19;99(4):584-90. doi: 10.1038/sj.bjc.6604536. Epub 2008 Jul 29. PMID 18665164
- [Background] O'Connell MJ, Laurie JA, Kahn M, Fitzgibbons RJ Jr, Erlichman C, Shepherd L, Moertel CG, Kocha WI, Pazdur R, Wieand HS, Rubin J, Vukov AM, Donohue JH, Krook JE, Figueredo A. Prospectively randomized trial of postoperative adjuvant chemotherapy in patients with high-risk colon cancer. J Clin Oncol. 1998 Jan;16(1):295-300. doi: 10.1200/JCO.1998.16.1.295. PMID 9440756
- [Background] Park JH, Ryu MH, Kim HJ, et al. (2012). Identification of risk factors of relapse after curative surgical resection in stage I gastric cancer. ESMO 2012 annual meeting, abstr number 679.
- [Background] Sakuramoto S, Sasako M, Yamaguchi T, Kinoshita T, Fujii M, Nashimoto A, Furukawa H, Nakajima T, Ohashi Y, Imamura H, Higashino M, Yamamura Y, Kurita A, Arai K; ACTS-GC Group. Adjuvant chemotherapy for gastric cancer with S-1, an oral fluoropyrimidine. N Engl J Med. 2007 Nov 1;357(18):1810-20. doi: 10.1056/NEJMoa072252. PMID 17978289
- [Background] Sasako M, Sakuramoto S, Katai H, Kinoshita T, Furukawa H, Yamaguchi T, Nashimoto A, Fujii M, Nakajima T, Ohashi Y. Five-year outcomes of a randomized phase III trial comparing adjuvant chemotherapy with S-1 versus surgery alone in stage II or III gastric cancer. J Clin Oncol. 2011 Nov 20;29(33):4387-93. doi: 10.1200/JCO.2011.36.5908. Epub 2011 Oct 17. PMID 22010012
- [Background] Lakatos E, Lan KK. A comparison of sample size methods for the logrank statistic. Stat Med. 1992 Jan 30;11(2):179-91. doi: 10.1002/sim.4780110205. PMID 1579757
- [Background] Collett, D. Modelling Survival Data in Medical Research, Chapman & Hall (1994), Section 9.2
- [Derived] Park JH, Ryu MH, Kim HJ, Ryoo BY, Yoo C, Park I, Park YS, Oh ST, Yook JH, Kim BS, Kang YK. Risk factors for selection of patients at high risk of recurrence or death after complete surgical resection in stage I gastric cancer. Gastric Cancer. 2016 Jan;19(1):226-33. doi: 10.1007/s10120-015-0464-5. Epub 2015 Jan 23. PMID 25614467